CLINICAL TRIAL: NCT04718285
Title: A National, Multi-Center, Open-Label, Three-Arm, Phase II Study to Investigate the Effect of Montelukast Between Emergency Room Visits and Hospitalizations in COVID-19 Pneumonia in Comparison With Standard Treatment
Brief Title: Investigation the Effect of Montelukast in COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bahçeşehir University (Other)
Collaborators: Medipol University (Other); The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Serdar Durdagi, Prof., Ph.D., Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MON786.168.1
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — montelukast; favipiravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Montelukast (Experimental): 3x10 mg oral montelukast first day (morning, noon time and evening) and rest of the 13 days 1 x 10 mg montelukast.
  Interventions: Drug: Montelukast Oral Tablet
- Montelukast plus Favicovir (Favipiravir) (Experimental): 200 mg oral favicovir for 5 days in a regimen of 2x1600 mg (oral) loading dose on day-1 (eight tablets in the morning and eight tablets in the evening) followed by 2x600 mg maintenance dose (three tablets in the morning and three tablets in the evening) on day-2 to day-5 and 3x10 mg oral montelukast at the first day and rest of the 13 days1 x 10 mg, concurrently.
  Interventions: Drug: Montelukast plus Favicovir (Favipiravir)
- Favicovir (Standard Treatment) (Active Comparator): 200 mg oral favicovir for 5 days in a regimen of 2x1600 mg (oral) loading dose on day-1 (eight tablets in the morning and eight tablets in the evening) followed by 2x600 mg maintenance dose (three tablets in the morning and three tablets in the evening) on day-2 to day-5.
  Interventions: Drug: Favicovir (Standard Treatment)

INTERVENTIONS:
Drug: Montelukast Oral Tablet — 3x10 mg oral montelukast first day and other 13 days 1 x 10 mg montelukast
  Arms: Montelukast
Drug: Montelukast plus Favicovir (Favipiravir) — 200 mg oral favicovir for 5 days in a regimen of 2x1600 mg (oral) loading dose on day-1 (eight tablets in the morning and eight tablets in the evening) followed by 2x600 mg maintenance dose (three tablets in the morning and three tablets in the evening) on day-2 to day-5 and 3x10 mg oral montelukast first day and rest of 13 days 1 x 10mg, concurrently.
  Arms: Montelukast plus Favicovir (Favipiravir)
Drug: Favicovir (Standard Treatment) — 200 mg oral favicovir for 5 days in a regimen of 2x1600 mg (oral) loading dose on day-1 (eight tablets in the morning and eight tablets in the evening) followed by 2x600 mg maintenance dose (three tablets in the morning and three tablets in the evening) on day-2 to day-5.
  Arms: Favicovir (Standard Treatment)

SUMMARY:
Small molecule inhibitors have previously been investigated in different studies as possible therapeutics in the treatment of SARS-CoV-2. In the current drug repurposing study, the investigators identified the leukotriene (D4) receptor antagonist Montelukast as a novel agent that simultaneously targets two important drug targets of SARS-CoV-2. The investigators initially demonstrated the dual inhibition (main protease and Spike/ACE2) profile of Montelukast through multiscale molecular modeling studies. Next, the investigators characterized its effect on both targets by different in vitro experiments including the Fluorescent Resonance Energy Transfer (FRET)-based main protease enzyme inhibition assay, surface plasmon resonance (SPR) spectroscopy, pseudovirus neutralization on HEK293T / hACE2, and virus neutralization assay using xCELLigence MP real time cell analyzer.

DETAILED DESCRIPTION:
The 2019 new coronavirus (SARS-CoV-2), was first reported in December 2019 in Wuhan (Hubei, China). It has quickly spread to other countries all around the world and effected more than 67 million people worldwide becoming an urgent global pandemic. Coronaviruses are enveloped, non-segmented positive-sense RNA viruses belonging to the family of Coronaviridae, the largest family in Nidovirales and widely distributed in humans, other mammals and birds, causing respiratory, enteric, hepatic and neurological diseases. Seven species of coronavirus are known to cause disease in humans. Four of them (229E, OC43, NL63, and HKU1) are common and they mostly cause common cold symptoms in immunocompetent individuals while the other three, SARS-CoV, MERS-CoV, and SARSCoV-2 cause serious symptoms and death.

SARS-CoV-2 has four structural proteins which are nucleocapsid, envelope, membrane and spike. These four proteins play a vital role during the viral infection. The Spike glycoprotein (S protein) located on the external surface of coronaviruses are responsible for the connection and entry of the virus to host cells. The S protein mediates receptor recognition, cell attachment, and fusion during viral infection. While the virus is in its natural environment, S protein of coronavirus is inactive. During viral infection, target cell proteases activate the S protein by cleaving it into S1 and S2 subunits, which are required to activate the membrane fusion domain after viral entry into target cells. The S1 subunit includes the receptor binding domain (RBD). This domain binds directly to the peptidase domain angiotensin converting enzyme 2 (ACE-2). S2 functions during membrane fusion. The chymotrypsin-like cysteine protease called 3C-like protease (3CLpro) aka main protease (Mpro) in SARS-CoV-2 is a vital enzyme involved in processes such as the processing, assembly, and replication of the virus.

One of the key characteristics of severe COVID-19 is increased cytokine production. It is thought that the severity of the disease is primarily associated with the cytokine storm, which is an aggressive immune response to the virus. The number of white blood cells, neutrophils, and levels of procalcitonin, C-reactive protein and other inflammatory indices like IL2, IL7, IL10, granulocyte-colony stimulating factor (GSCF), interferon inducible protein -10 (IP10), monocyte chemotactic protein-1 (MCP1), macrophage inflammatory protein-1α (MIP1A), and TNF are significantly higher in severe cases in patients with COVID-19. Specifically, IL-1β, IL-6, and IL-10 are the three most elevated cytokines in serious cases. One result of the cytokine storm is lung injury that can develop into acute lung injury or its more severe type (acute respiratory distress syndrome, ARDS). Studies have shown the relation between COVID-19 and the most common chronic conditions such as diabetes, cardiovascular diseases, respiratory system diseases, immune system disorders, etc. Asthma and chronic obstructive pulmonary disease (COPD) are among the diseases of the respiratory system that are most emphasized. Asthma is a chronic inflammatory airway condition. There is significant evidence that represents the relation of asthmatic patients in the population with viral infections like rhinoviruses. Virus infections cause upper respiratory tract infection, like influenza A, rhinovirus, and respiratory syncytial virus (RSV) elevate local leukotriene levels. Leukotrienes, which play a role in the contraction of bronchial muscles, are effective in initiating and amplifying many biological responses, including mast cell cytokine secretion, macrophage activation, and dendritic cell maturation and migration. Leukotrienes (LTC4, LTD4 and LTE4), activated basophils, eosinophils, macrophages, and products of mast cells are types of lipids conjugated with peptides. LTD4 receptors belong to G protein-coupled receptor (GPCR) family. Montelukast is a selective leukotriene (D4) receptor antagonist which is a member of quinolines and it was approved by FDA as an oral tablet in 1998. It is a licensed drug used for allergic rhinitis, exercise-induced bronchospasm and especially prophylaxis and chronic treatment of asthma. As a result of LTD4 blockage, NF-kB pathway activation and release of the proinflammatory mediators (i.e., IL-6,8 and 10, TNF-a and MCP-1) decrease. Considering these anti-inflammatory effects by leukotriene receptor inhibition and possible antiviral effects, Montelukast maybe considered for the effective medication against SARS CoV-2.

Here, initially the investigators explored the potential role of Montelukast in the management of SARS-CoV-2 infection with multiscale molecular modeling approaches and its promising results both in main protease and Spike/ACE2 interface encouraged the investigators to perform further detailed in vitro experiments. The results of FRET-based biochemical assays, surface plasmon resonance (SPR), pseudovirus neutralization and virus neutralization experiments demonstrated the effect of Montelukast on SARS-CoV-2.

This study was designed as a national, multi-center, open-label, randomized, parallel, three-arm, phase-II study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years and older infected with the SARS-CoV-2 infection
* Patients with COVID-19 symptoms and have a positive PCR test result
* Patients in a stable clinical condition and basically in an outpatient condition
* Patients who sign the informed consent

Exclusion Criteria:

* Patients with a partial oxygen pressure < 90% and who have required hospitalization
* Patients who have required intensive care
* Any condition which, in the opinion of the Principal Investigator, would prevent full participation in and compliance with the trial protocol
* Patients who have been involved in any other interventional studies
* Patients with uncontrolled Type I or Type II diabetes mellitus (DM)
* Patients with severe liver failure (Child Pugh score ≥ C, AST> 5 times the upper limit of normal (ULN)
* Patients with severe renal failure (GFR ≤30 mL/min/1.73 m2) or continuous dialysis (hemodialysis, peritoneal dialysis) or continuous renal replacement therapy
* Patients with serious cardiac problems such as heart failure
* Patients with hypersensitivity to montelukast or other drugs in the study
* Patients with rare hereditary problems of galactose / fructose intolerance, glucose- galactose malabsorption or sucrase-isomaltase insufficiency
* Pregnant and lactating women
* Patients who cannot use sexual abstinence or appropriate contraceptive method during the study
* Patients who are treated with any other antiviral drugs for COVID-19 in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Hospitalized patient rates | 15 days
  The number of hospitalized patients

SECONDARY OUTCOMES:
Emergency room visit rates of patients | 15 days
  The number of emergency room visits of patients not hospitalized
Time to emergency room visit | 15 days
  The time (days) until the emergency room visit
Time to hospitalization | 15 days
  The time (days) until the hospitalization
Inpatient length of stay | 15 days
  Length of stay in the hospital (days)
Time to ICU admission | 15 days
  The time (days) until admission to intensive care unit
Time to intubation | 15 days
  The time (days) until intubation
Mortality rate | 15 days
  All-cause mortality rate
Family members rates with PCR positive test results | 15 days
  The number of family members with PCR positive
Number/characteristics of AEs and SAEs | 21 days
  Number/characteristics of Adverse Event (AE) and Serious Adverse Event (SAE) related to study drug or hematological and biochemical parameters from baseline until the end of study
Changes in blood pressure from baseline | 21 days
  Clinical evaluation of systolic and diastolic blood pressure changes from baseline until the end of study
Changes in pulse from baseline | 21 days
  Clinical evaluation of pulse values from baseline until the end of study
Changes in respiratory rate from baseline | 21 days
  Clinical evaluation of respiratory rate levels from baseline until the end of study
Changes in fever from baseline | 21 days
  Clinical evaluation of fever changes from baseline until the end of study
Changes in oxygen saturation from baseline | 21 days
  Clinical evaluation of oxygen saturation changes from baseline until the end of study

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bahcesehir University, School of Medicine, Department of Biophysics,, Istanbul
  - Istanbul University, Cerrahpaşa School of Medicine, Istanbul

REFERENCES:
- [Background] Durdagi S, Avsar T, Orhan MD, Serhatli M, Balcioglu BK, Ozturk HU, Kayabolen A, Cetin Y, Aydinlik S, Bagci-Onder T, Tekin S, Demirci H, Guzel M, Akdemir A, Calis S, Oktay L, Tolu I, Butun YE, Erdemoglu E, Olkan A, Tokay N, Isik S, Ozcan A, Acar E, Buyukkilic S, Yumak Y. The neutralization effect of montelukast on SARS-CoV-2 is shown by multiscale in silico simulations and combined in vitro studies. Mol Ther. 2022 Feb 2;30(2):963-974. doi: 10.1016/j.ymthe.2021.10.014. Epub 2021 Oct 19. PMID 34678509